CLINICAL TRIAL: NCT06640777
Title: Multicenter, Randomized, Open-Label Phase 3 Study to Investigate Efficacy and Safety of Liposomal Transcrocetin(LEAF-4L6715) Plus Standard of Care Vs Standard of Care Alone for Treatment of Patients with Acute Respiratory Distress Syndrome
Brief Title: Efficacy and Safety of LEAF-4L6715 for Acute Respiratory Distress Syndrome
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: LEAF4Life, Inc. (Industry)
Collaborators: European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEAF-4L6715-03-01-01
Record Dates: First submitted 2024-08-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-08

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: Prospective, international, multicenter, open label, randomized, controlled, two-arm study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LEAF-4L6715 (Liposomal Transcrocetin) + Supportive Care (Experimental): LEAF-4L6715 administered Intravenously 200 mg every 12h for 2 days, then 200 mg Intravenously every 24 hours for 8 days (total 10 days dosing)
  Supportive care, as considered necessary by the treating physician/Principal Investigator (PI), including mechanical ventilation, in line with therapeutic guidelines for ARDS and Multiorgan Failure
  Interventions: Drug: LEAF-4L6715; Drug: Supportive Care
- Supportive Care (Active Comparator): Description: Supportive care, as considered necessary by the treating physician/Principal Investigator (PI), including mechanical ventilation, in line with therapeutic guidelines for ARDS and Multiorgan Failure
  Interventions: Drug: Supportive Care

INTERVENTIONS:
Drug: LEAF-4L6715 — LEAF-4L6715: Administration at a dose of 200mg , for up to 10 days every 12 hours for the first 2 days, followed by once-a-day dosing for the next 8 days (days 3 through 10).
  Other Names: Liposomal transcrocetin
  Arms: LEAF-4L6715 (Liposomal Transcrocetin) + Supportive Care
Drug: Supportive Care — Supportive care, as considered necessary by the treating physician/Principal Investigator (PI), including mechanical ventilation, in line with therapeutic guidelines for ARDS and Multiorgan Failure

SUMMARY:
Acute Respiratory Distress Syndrome (ARDS) is a serious condition where people in hospital care suddenly have trouble breathing because of infection, pneumonia, COVID-19 or other disease. People with ARDS may have to be put in an intensive care unit (ICU) and on a ventilator to help them breathe. This trial is to try to find out if injecting a product called LEAF-4L6715 makes the treatment better or worse than what is normally given. LEAF-4L6715 is a product that contains tiny bubbles to slowly release a substance named transcrocetin which scientific studies show may increase oxygen flow and reduce inflamed cells and protect tissues of the body.

DETAILED DESCRIPTION:
Study Design: Prospective, international, multicenter, open label, randomized, controlled, two-arm study.

Study Objective(s): The primary objective of the study is to determine if the addition of LEAF-4L6715 to Standard of Care (SOC) treatment may improve clinical outcomes at 30-days, including survival and duration of mechanical ventilation (MV), in patients with Acute Respiratory Distress Syndrome (ARDS) compared to SOC treatment alone.

The secondary objectives are to compare other relevant respiratory and clinical outcomes and safety between the two groups during Intensive Care Unit (ICU) stay, hospitalization, and follow-up, including percentage of patients alive at 60 days and 90 days from randomization.

Rationale: The scientific and clinical observations to date strongly suggest that transcrocetin (TC) may be a good candidate for the treatment of hypoxic conditions such as moderate to severe ARDS. Indeed, TC plays a major role in enhancing oxygen diffusion, but also in reducing inflammation and protecting tissues. However, TC's poor stability and solubility and its short in vivo half-life of ~30mins resulted in transient oxygenation effect. LEAF-4L6715 was designed to be a stable TC formulation with a 6-fold increase in half-life and a 12-fold increase in drug exposure compared to free TC, resulting in a more sustained oxygenation compared with free TC.

Developed as a liposomal formulation of TC, LEAF-4L6715 allows for a gradual release of the free drug and was evaluated at multiple levels (1) in vitro in Human Umbilical Vein Endothelial Cells (HUVECs); (2) in vivo in healthy mice (n=40) as well as in a mouse model of sepsis (n=10) and (3) in a clinical trial evaluating Pharmacokinetics (PK) and safety. A phase 1/2 trial which included 37 patients defined the optimal dose regimen and intravenous infusion timing and confirmed the safety of LEAF-4L6715. It also showed promising trends in therapeutic efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if all of the following criteria are met:

  1. Patients ≥18 years old
  2. Signed and dated informed consent from patient's trusted person before any study related procedures, pursuing patient signature as soon as patient health condition allows
  3. ARDS with a documented Positive End-Expiratory Pressure (PEEP) ≥5 and PaO2/FiO2 ratio of ≤200 mm Hg for a minimum of 24 hours prior to randomization
  4. Patient with an endotracheal tube or tracheostomy tube and receiving MV support
  5. Life expectancy of at least 24 hours from randomization
  6. Alanine transaminase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP) < 3 x upper limit of normal at the time of randomization
  7. Male or non-pregnant female patient
  8. Affiliated to a social security system (for France)

Exclusion Criteria:

1. Enrolled in any other therapeutic clinical trial or receiving an experimental drug (only observational studies allowed)
2. Hypersensitivity to crocetins, LEAF 4L6715 or any of its excipients.
3. Receiving extracorporeal membrane oxygenation (ECMO) treatment
4. On MV for more than 7 days
5. Chronic Obstructive Pulmonary Disease (COPD) or other respiratory insufficiency with home ventilation or oxygen therapy
6. Severe underlying pre-existing condition with expected 6 months mortality >50% or survival <50%
7. Patient moribund, decision to limit therapeutic interventions
8. Unwilling or unable to comply with study procedures
9. Under guardianship, curatorship or safeguard of justice (for France)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-11-09 (Estimated); Study Completion 2027-11-09 (Estimated)

PRIMARY OUTCOMES:
Days free from invasive mechanical ventilation | 30 Days
  From Randomization to Day 30
30 Day All-Cause Mortality | 30 days
  Survival at Day 30

SECONDARY OUTCOMES:
Mean total of Sequential Organ Failure Assessment (SOFA) score | 30 days
  Mean total of Sequential Organ Failure Assessment (SOFA) score and sub-scores during the treatment period.
Need for rescue procedures | 30 days
  Need for rescue procedures such as prone positioning, inhaled nitric oxide (NO), recruitment maneuvers, extracorporeal membrane oxygenation (ECMO).
Ventilator-associated pneumonia treated with antibiotics between randomization and 30 days. | 30 days
  Proportion of patients with ventilator-associated pneumonia treated with antibiotics between randomization and 30 days.
Number of days alive without organ failure at 30 days and 60 days | 60 days
  Number of days alive without organ failure at 30 days and 60 days, using the SOFA score and its components
Mean reduction in the WHO 9-point Ordinal Scale score | 30 days
  Mean reduction in the WHO 9-point Ordinal Scale score from start of treatment to 30 days
Length of ICU stay | 60 days
  Number of days patient was in Intensive Care Unit
Length of hospital stay | 60 Days
  Number of days patient stayed in hospital
Incidence of serious adverse events (SAEs), AEs, and treatment-emergent adverse events | 90 Days or event resolution/stabilization
  Incidence of serious adverse events (SAEs), AEs, and treatment-emergent adverse events by maximum Common Terminology Criteria for Adverse Events (CTCAE) grade and/or change in baseline laboratory values
Change in Quality of Life (QOL) by Health economics and outcomes research assessments | 90 days
  Change in Quality of Life (QOL) by Health economics and outcomes research assessments: to compare patient QOL using European QOL Five Dimension (EQ-5D-5L)
Survival at 30, 60 and 90 days | 90 days
  Number of patients alive at 30, 60 and 90 days from randomization.
PaO2/FiO2 ratio | 30 days
  Number of patients with an improvement of 25% in PaO2/FiO2 ratio at 72 hours post-treatment initiation and over time until acute treatment discontinuation.
Time to successful extubation | 30 days
  Time in hours to successful extubation without re-intubation or death within the next 48 Hours
Total duration of mechanical ventilation | 30 days
  Total duration of MV in days and the number of days, between randomization and 30 days, alive without MV.
Pharmacokinetics (PK) assessments | Day 1, Day 3, Day 14 and Day 30
  12. Maximum plasma concentration (Cmax) , units μg/ml
Pharmacokinetic (PK) Assessments | Day 1, Day 3, Day 14 and Day 30
  Area under the curve (AUC) units h*μg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Alain Combes, MD, Principal Investigator — Hôpital de la Pitié Salpêtrière; Marie Claude Morice, Ph.D., Study Director — CERC - CARDIOVASCULAR EUROPEAN RESEARCH CENTER; Clet Niyikiza, Ph.D., Study Chair — LEAF4Life, Inc.
Locations (1):
- Sorbonne University, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No